CLINICAL TRIAL: NCT04826822
Title: Spironolactone and Dexamethasone in Patients Hospitalized With Moderate-to-severe COVID-19 (SPIDEX-II): a Randomized Clinical Trial
Brief Title: Spironolactone and Dexamethasone in Patients Hospitalized With COVID-19
Acronym: SPIDEX-II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chita State Regional Clinical Hospital Number 1 (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPII_1789461
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infection; Pneumonia, Viral
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral | interventions — Spironolactone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): After randomisation (Day 1): Spironolactone [100 mg 1x/day] + dexamethasone [2 mg 2x/day, 12/12h] Days 2-12*: Spironolactone [50 mg 2x/day, 12/12h] + dexamethasone [2 mg 2x/day, 12/12h] Days 13-20: Spironolactone [25 mg 2x/day, 12/12h] Days 21-28: Spironolactone [25 mg 1x/day] Standard treatment is according to the treatment protocol for 2019-nCoV infection.
  *In case of cortisol levels above 100 nmol/L on days 3 and 4, the dexamethasone dose should be increased to 3 mg in the morning and in the evening (total 6 mg per day).
  Interventions: Drug: Spironolactone + Dexamethasone
- Control (Active Comparator): Patients receiving standard-of-care treatment for SARS-CoV-2 infection as regulated by the relevant guidelines of the Ministry of Healthcare of the Russian Federation
  Interventions: Drug: Standard-of-care SARS-CoV-2 treatment

INTERVENTIONS:
Drug: Spironolactone + Dexamethasone — Low doses of orally administered spironolactone and dexamethasone
  Arms: Treatment
Drug: Standard-of-care SARS-CoV-2 treatment — Standard-of-care SARS-CoV-2 treatment administered according to the local guidelines
  Arms: Control

SUMMARY:
The Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) is a rapidly spreading infection of the respiratory tract. Most infected patients have either asymptomatic disease or mild symptoms. However, a proportion of patients, especially elderly men or patients with comorbidities, are at risk of developing acute respiratory distress syndrome (ARDS). ARDS, alongside clotting abnormalities, is known to be a major contributor to SARS-CoV-2-related mortality and admission to intensive care units, with evidenced effective preventative treatment options lacking. In this study, the investigators test a novel hypothesis that the use of a combination of spironolactone and dexamethasone at low doses will improve the clinical progression of the infection evaluated by the 6-point ordinal scale in patients with moderate and severe disease by blocking exocytosis of the Weibel-Palade bodies from endothelial cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above;
* Signed informed consent;
* PCR-confirmed diagnosis of SARS-CoV-2 infection
* Presenting with moderate-to-severe disease (scores 4-6 on WHO ordinal scale)

Exclusion Criteria:

* Women of childbearing age without a negative urine pregnancy test, currently pregnant or breastfeeding women;
* Severe heart failure (NYHA4), severe renal failure (eGFR < 30 ml/min/1.73 m2), severe liver failure (ALT/AST ratio > 5 norms), severe anemia (haemoglobin < 30 g/l)
* Participating in another clinical trial
* Severe electrolyte imbalance (hyperkalemia > 5.0 mmol/l, hyponatremia < 120 mmol/l)
* Hypersensitivity or contraindications to the study drugs (spironolactone and dexamethasone)
* Renal dialysis
* Severe uncontrolled diabetes mellitus
* Patient receiving one of the following medications that cannot be substituted over the trial duration: ACE inhibitors, amiloride, eplerenone, cortisone acetate, potassium canrenoate, triamterene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-07-08 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the clinical status | Day 14 post-randomization
  Clinical status at day 14 post-randomization defined by a 6-point ordinal scale score (6 being the worst score)

SECONDARY OUTCOMES:
28-day all-cause mortality | 28 days post-randomization
  All-cause mortality at 28 days post-randomization
Oxygen-free days | 28 days post-randomization
  The number of days without oxygen support of any type
Ventilator-free days | 28 days post-randomization
  The number of days without invasive mechanical ventilation
Invasive mechanical ventilation | 28 days post-randomization
  The number of patients requiring invasive mechanical ventilation during hospitalization and the number of days spent on newly-administered invasive mechanical ventilation
Time to discharge | 28 days post-randomization
  The number of days from hospitalization to discharge
Length of ICU stay | 28 days post-randomization
  The number of days spent in the intensive care unit
New ICU admission | 28 days post-randomization
  The number of patients requiring transfer to ICU and the number of days spent in the ICU post-transfer
Long-COVID development | 60 and 90 days post-admission
  The number of patients with signs and symptoms that develop during or after an infection consistent with COVID-19, continue for more than 12 weeks and are not explained by an alternative diagnosis (Post-COVID-19 syndrome as defined by the relevant NICE guidance)
Evaluation of the clinical status | Day 7 post-randomization
  Clinical status at day 7 post-randomization defined by a 6-point ordinal scale score (6 being the worst score)

OTHER OUTCOMES:
Adverse events | 28 days post-randomization
  Incidence of adverse events related to the use of the investigational products
Laboratory abnormalities | 28 days post-randomization
  Occurrence of laboratory hematimetric parameters, creatinine, d-dimer, c-reactive protein
Change in classic cough score | 28 days post-randomization
  Change in classic cough score measured daily in hospitalized patients
Radiological abnormalities | 28 days post-randomization
  Occurrence of viral pneumonia-associated changes on sequential chest CT scans in hospitalized patients

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Lukyanov, MD, Principal Investigator — Chita State Regional Clinical Hospital Number 1
Locations (1):
- Chita State Regional Clinical Hospital Number 1, Chita, Russia

IPD SHARING:
Plan to Share IPD: No
Sharing IPD would require material transfer agreement according to the local rules and regulations. The study protocol, statistical analysis plan, and the translated version of the informed consent form can be shared upon request.